CLINICAL TRIAL: NCT05146479
Title: A Long-term Retrospective Cohort Study in Children With Autism Spectrum Disorders on the Effectiveness of Dental Sealants and Fluoride Varnish to Prevent the Occurrence of New Caries
Brief Title: Effectiveness of Sealants and Fluoride Varnish in Caries Prevention in Children With Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Maria Grazia Cagetti, Prof. Maria Grazia Cagetti, University of Milan
Other Study IDs: 0000546
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Autistic Disorder; Dental Caries; Pit and Fissure Caries
Keywords: Dental sealant; Pit and Fissure sealant; Preventive dentistry; Fluoride varnish
MeSH Terms: conditions — Autistic Disorder; Dental Caries; Van der Woude syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fluoride varnish (FA group): Application of 5% NaF varnish onto first permanent molars
- Fluoride varnish + dental sealant (FA+S group): Application of 5% NaF varnish plus pit and fissure sealant onto first permanent molars
  Interventions: Procedure: Fluoride varnish and pit and fissure sealants onto first permanent molars

INTERVENTIONS:
Procedure: Fluoride varnish and pit and fissure sealants onto first permanent molars — Quarterly application of fluoride varnish. Application of pit and fissure sealant, and replacements if necessary.
  Groups: Fluoride varnish + dental sealant (FA+S group)

SUMMARY:
The aim of the study is to compare application of sealants together with fluoride varnishes versus only fluoride varnishes in preventing caries lesions development in the occlusal surface of first permanent molars of children with ASDs.

DETAILED DESCRIPTION:
The aim of the study is to evaluate if the application of pit and fissure sealants together with fluoride varnishes is more effective than the application of the only fluoride varnishes in preventing caries lesions development in the occlusal surface of first permanent molars of children with ASDs.

Patients with at least 10-year follow-up and ASDs are recruited and allocated to two cohort according to the strategy adopted for prevention of caries in first permanent molars: FA group (only fluoride varnishes) and FA+S group (sealants together with fluoride varnishes).

Caries incidence and sealants retention after the follow-up period are recorded. Demographic and clinical characteristics of patients at first dental visit are also recorded (age, level of cooperation, presence of systemic diseases other than ASDs, caries severity) to evaluate if they play a potential protective and/or risk factors for caries development.

Logistic and multivariate analysis are run to evaluate caries incidence and retention rate of sealants in first permanent molars over a period of at least 10 years.

ELIGIBILITY:
Inclusion Criteria:

* ASDs
* age less than 14 years
* written declaration of informed consent signed by parents/guardians

Exclusion Criteria:

* incomplete clinical records
* missing five or more dental check-ups over the follow-up period
* oral or dental care provided in sedation or general anesthesia
* follow-up less than 15 years

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary care clinic: participants were enrolled among those who have being received dental care at the Dental Service for ASD children of San Paolo Hospital, Milan, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Survival rates from dental caries | 15 years
  Percentage of first permanent molars free from caries

SECONDARY OUTCOMES:
Survival rates of pit and fissure sealant | 15 years
  Percentage of pit and fissure sealant sound
Evaluation of confounders | 15 years
  Evaluation if patient's variables at the first dental visit, such as age, number of dental caries, cooperation level, are positively or negatively associated with first permanent molars decay rates overtime.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia MG Cagetti, Prof, Study Chair — University of Milan
Locations (1):
- Dental Clinic San Paolo Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request